CLINICAL TRIAL: NCT05247164
Title: EUS-guided PORtal Vein Sampling for Isolation, Enumeration and Profiling of Circulating Tumor Cells in Pancreatic Cancer Patients
Brief Title: EUS-guided PORtal Vein Sampling for Circulating Tumor Cells in Pancreatic Cancer Patients
Acronym: EUPhORIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giuseppe Vanella, Principal Investigator, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 129/INT/2021
Record Dates: First submitted 2022-02-06; First posted 2022-02-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: Endoscopic Ultrasound; EUS; Portal blood; Circulating Tumor Cells; Fine Needle Aspiration
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDAC Patients (Experimental): Patients undergoing EUS for characterization of a PDAC lesion will receive EUS-guided portal blood sampling.
  Interventions: Procedure: EUS-guided Portal Vein sampling

INTERVENTIONS:
Procedure: EUS-guided Portal Vein sampling — Transgastric and Transhepatic Fine Needle Aspiration of a branch of the Portal Vein under EUS guidance.
  A paired peripheral sample will be acquired.

SUMMARY:
The study aims at evaluating the feasibility and safety of EUS-guided Portal Circulation sampling for isolation, enumeration and profiling od Circulating Tumor Cells (CTC) in Pancreatic Cancer patients.

Patients undergoing Endoscopic Ultrasound (EUS) for cyto/histological characterization of the neoplasia will receive an additional Fine Needle Aspiration sampling of a branch of the Portal Circulation to obtain a blood sample which will be processed for CTC enrichment, count and characterization.

DETAILED DESCRIPTION:
Prognostic stratification of patients with Pancreatic Ductal Adenocarcinoma (PDAC) is still suboptimal, relying only on imaging studies and Carbohydrate Antigen 19.9 to drive important treatment decisions (e.g. surgery versus neoadjuvant chemotherapy).

Circulating Tumor Cells (CTCs) have been poorly evaluated in this neoplasia as they are rarely detected in the peripheral blood, whereas they are more abundantly detected in the portal circulation below the hepatic filter.

Most PDAC patients undergo Endoscopic Ultrasound (EUS) for cyto/histological characterization of the neoplasia. EUS-guided acquisition of portal blood for CTC evaluation has demonstrated its feasibility in preliminary studies without reducing the safety of the endoscopic procedure.

The study aims at collecting portal blood from PDAC patients under EUS-guidance to evaluate whether concentration and characterization of CTCs has a prognostic significance and can aid in decision making.

A paired peripheral blood sample will be acquired for comparison. Samples will be processed to obtain microfluidic enrichment of CTCs and stained with immunofluorescent antibodies for exclusion of hematopoietic cells and specific identification of CTCs, which will then be counted to obtain the blood concentration expressed as number of cells per 7.5 ml of blood.

Patients will be followed every 60 days for a maximum of 24 months to assess the evolution of primary disease and clinical status.

ELIGIBILITY:
Inclusion Criteria:

* patient with a pancreatic solid lesion undergoing EUS with a rapid on-site confirmation of a pancreatic ductal adenocarcinoma
* patients primarily followed within San Raffaele Institute

Exclusion Criteria:

* history of active non-pancreatic cancer
* coagulopathy (INR > 1.5; platelets < 70.000/ul) or use of non-withdrawable anticoagulant or antiplatelet
* known history or endosonographic signs of portal hypertension
* extensive invasion of portal vein precluding needle maneuvers
* pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with successful aspiration of portal blood | Day 1
  The proportion of patients with successful needle access to the portal circulation with subsequent successful aspiration of portal blood
Proportion of patients with procedure-related Adverse Events | 30 days
  The proportion of patients experiencing procedure-related adverse events, such as bleeding or perihepatic collections.

SECONDARY OUTCOMES:
Difference between Portal and Peripheral CTC concentration | Day 1
  CTC concentration [Count / 7.5 ml of blood]
Portal CTC concentration according to clinical stage | Day 1
  CTC concentration [Count / 7.5 ml of blood]
Baseline portal CTC concentration in patients with progressive versus non-progressive diseases | 24 months
  CTC concentration [Count / 7.5 ml of blood]

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Vanella, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catenacci DV, Chapman CG, Xu P, Koons A, Konda VJ, Siddiqui UD, Waxman I. Acquisition of Portal Venous Circulating Tumor Cells From Patients With Pancreaticobiliary Cancers by Endoscopic Ultrasound. Gastroenterology. 2015 Dec;149(7):1794-1803.e4. doi: 10.1053/j.gastro.2015.08.050. Epub 2015 Sep 2. PMID 26341722
- [Background] Liu X, Li C, Li J, Yu T, Zhou G, Cheng J, Li G, Zhou Y, Lou W, Wang X, Gong G, Liu L, Chen Y. Detection of CTCs in portal vein was associated with intrahepatic metastases and prognosis in patients with advanced pancreatic cancer. J Cancer. 2018 May 22;9(11):2038-2045. doi: 10.7150/jca.23989. eCollection 2018. PMID 29896289
- [Background] Pang TCY, Po JW, Becker TM, Goldstein D, Pirola RC, Wilson JS, Apte MV. Circulating tumour cells in pancreatic cancer: A systematic review and meta-analysis of clinicopathological implications. Pancreatology. 2021 Jan;21(1):103-114. doi: 10.1016/j.pan.2020.11.022. Epub 2020 Dec 3. PMID 33309014
- [Background] Zhang Y, Su H, Wang H, Xu C, Zhou S, Zhao J, Shen S, Xu G, Wang L, Zou X, Zhang S, Lv Y. Endoscopic Ultrasound-Guided Acquisition of Portal Venous Circulating Tumor Cells as a Potential Diagnostic and Prognostic Tool for Pancreatic Cancer. Cancer Manag Res. 2021 Oct 5;13:7649-7661. doi: 10.2147/CMAR.S330473. eCollection 2021. PMID 34675662